CLINICAL TRIAL: NCT05494320
Title: The Effect of ATP-Binding Cassette C2 (ABCC2) Transporter Genetic Polymorphism on Neurotoxicity in Gastrointestinal Cancer Patients Receiving Oxaliplatin -Based Chemotherapy
Brief Title: the Effect of ABCC2 Genetic Polymorphism on Neurotoxicity in Gastrointestinal Cancer Patients Receiving Oxaliplatin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Abdel Aziz Mohamed, pharmacist, Ain Shams University
Other Study IDs: 279
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Gastrointestinal Cancer
Keywords: neurotoxicity; oxaliplatin; genetic polymorphism
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neurotoxicity Syndromes | interventions — Folfox protocol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Folfox Protocol — Folfox: It includes the drugs leucovorin calcium (folinic acid), fluorouracil, and oxaliplatin.
  Other Names: Folfox_6

SUMMARY:
Study the effect of genetic polymorphism (rs1885301, rs4148396 and rs3740066) in the membrane of Multidrug resistance protein 2 (MRP2) encoded by ATP-binding cassette C2 (ABCC2) gene and its genetic expression levels on neurotoxicity in gasrtointestinal cancer patients reciving Oxaliplatin-based chemotherapy.

DETAILED DESCRIPTION:
Several solutes carriers and ATP-binding cassette transporters have been implicated in the influx or efflux of platinum-based chemotherapeutic agents such as cisplatin, carboplatin, and oxaliplatin. The ATP-binding cassette (ABC-) transporter superfamily contains several family members that may confer intrinsic or acquired multidrug resistance (MDR) by extruding anticancer agents or their metabolites from cells and suppression of such transporters may lead to sensitisation to cytostatic agents. Multidrug resistance protein 2 (MRP2), encoded by the ATP-binding cassette C2 (ABCC2) gene , is an efflux pump located on the apical membrane of many polarized cells, which transports conjugate compounds by an ATP-dependent mechanism like oxaliplatin. Single nucleotide polymorphisms (SNPs) in genes involved in drug transport like ABCC2 gene may lead to higher intracellular oxaliplatin accumulation in the dorsal root ganglia and thus increased risk of Oxaliplatin-induced peripheral neurotoxicity (OXPN). Enhanced ABCC2 expression can lead to decreased cellular glutathione content. Glutathione is needed for oxaliplatin detoxification via conjugation, and it was reported that low glutathione intra- cellular levels can cause increased oxaliplatin cytotoxicity. Moreover, ABCC2 mediates the export of the oxaliplatin-glutathione conjugated form, and ABCC2 overexpressing cells were resistant to platinum derivatives.

ELIGIBILITY:
Inclusion Criteria:

1. gastrointestinal cancer Patients ( ≥ stages II ) who receive Oxaliplatin based chemotherapy ( FOLFOX6 ) for adjuvant and metastatic setting.
2. Eastern Cooperative Oncology Group ( ECOG ) performance ≤ 2.
3. Adequate bone marrow functions ,liver functions and renal functions.

Exclusion Criteria:

1. Patients who have any clinical neuropathy.
2. Pateints with Diabetes mellitus.
3. Serious comorbid systemic disorder incompatible with study.
4. Pregnancy.
5. Other primary tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the pateints presenting to the department of Clinical Oncology Department, Ain Shams University Hospitals with gastrointestinal cancer (stage ≥ stages II ) who receive Oxaliplatin based chemotherapy ( FOLFOX6 ) for adjuvant and metastatic setting.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
neurotoxicity | 6 months
  the effect of genetic polymorphism (rs1885301, rs4148396 and rs3740066) in the membrane of Multidrug resistance protein 2 (MRP2) encoded by ATP-binding cassette C2 (ABCC2) gene and its genetic expression levels on neurotoxicity in gastrointestinal cancer patients reciving Oxaliplatin-based chemotherapy.
  Grading of peripheral neuropathy using National Cancer Institute's Common Toxicity Criteria for Adverse Event ( NCI- CTCAE V5.0 ) will be assessed at baseline and before each cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Ali Sabri, Professor, Study Director — Clinical Pharmacy Department - Faculty of Pharmacy - Ain Shams University; May Ahmed Shawki, Lecturer, Study Director — Clinical Pharmacy Department - Faculty of Pharmacy - Ain Shams University; Diaa Eldin Moussa Sherif, Lecturer, Study Director — Clinical oncology and nuclear medicine Department -Faculty of medicine-Ain Shams University; Sara Mohamed Abdel Aziz, Master Student, Principal Investigator — Clinical Pharmacy Department - Faculty of Pharmacy - Ain Shams University
Locations (1):
- Ain shams university, Cairo, Abassia, Egypt

REFERENCES:
- [Background] Alberti P, Rossi E, Cornblath DR, Merkies IS, Postma TJ, Frigeni B, Bruna J, Velasco R, Argyriou AA, Kalofonos HP, Psimaras D, Ricard D, Pace A, Galie E, Briani C, Dalla Torre C, Faber CG, Lalisang RI, Boogerd W, Brandsma D, Koeppen S, Hense J, Storey D, Kerrigan S, Schenone A, Fabbri S, Valsecchi MG, Cavaletti G; CI-PeriNomS Group. Physician-assessed and patient-reported outcome measures in chemotherapy-induced sensory peripheral neurotoxicity: two sides of the same coin. Ann Oncol. 2014 Jan;25(1):257-64. doi: 10.1093/annonc/mdt409. Epub 2013 Nov 19. PMID 24256846
- [Background] Andre T, Boni C, Navarro M, Tabernero J, Hickish T, Topham C, Bonetti A, Clingan P, Bridgewater J, Rivera F, de Gramont A. Improved overall survival with oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment in stage II or III colon cancer in the MOSAIC trial. J Clin Oncol. 2009 Jul 1;27(19):3109-16. doi: 10.1200/JCO.2008.20.6771. Epub 2009 May 18. PMID 19451431
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Cappell MS. Pathophysiology, clinical presentation, and management of colon cancer. Gastroenterol Clin North Am. 2008 Mar;37(1):1-24, v. doi: 10.1016/j.gtc.2007.12.002. PMID 18313537
- [Background] Cecchin E, D'Andrea M, Lonardi S, Zanusso C, Pella N, Errante D, De Mattia E, Polesel J, Innocenti F, Toffoli G. A prospective validation pharmacogenomic study in the adjuvant setting of colorectal cancer patients treated with the 5-fluorouracil/leucovorin/oxaliplatin (FOLFOX4) regimen. Pharmacogenomics J. 2013 Oct;13(5):403-9. doi: 10.1038/tpj.2012.31. Epub 2012 Aug 7. PMID 22868256
- [Background] Ewertz M, Qvortrup C, Eckhoff L. Chemotherapy-induced peripheral neuropathy in patients treated with taxanes and platinum derivatives. Acta Oncol. 2015 May;54(5):587-91. doi: 10.3109/0284186X.2014.995775. Epub 2015 Mar 9. PMID 25751757
- [Background] Grady WM, Markowitz SD. The molecular pathogenesis of colorectal cancer and its potential application to colorectal cancer screening. Dig Dis Sci. 2015 Mar;60(3):762-72. doi: 10.1007/s10620-014-3444-4. Epub 2014 Dec 10. PMID 25492499
- [Background] Nichetti F, Falvella FS, Miceli R, Cheli S, Gaetano R, Fuca G, Infante G, Martinetti A, Antoniotti C, Falcone A, Di Bartolomeo M, Cremolini C, de Braud F, Pietrantonio F. Is a pharmacogenomic panel useful to estimate the risk of oxaliplatin-related neurotoxicity in colorectal cancer patients? Pharmacogenomics J. 2019 Oct;19(5):465-472. doi: 10.1038/s41397-019-0078-0. Epub 2019 Feb 4. PMID 30713338
- [Background] Mirakhorli M, Rahman SA, Abdullah S, Vakili M, Rozafzon R, Khoshzaban A. Multidrug resistance protein 2 genetic polymorphism and colorectal cancer recurrence in patients receiving adjuvant FOLFOX-4 chemotherapy. Mol Med Rep. 2013 Feb;7(2):613-7. doi: 10.3892/mmr.2012.1226. Epub 2012 Dec 7. PMID 23232902
- [Background] Nguyen TQ, Bui TO, Tran PT, Tran VT, Nguyen VH, Chu QH, Bui TAT, Le NQ, Le VQ, Dao VT. Modified Folfox6 as Adjuvant Chemotherapy in Vietnamese Patients With Colorectal Cancer. Cancer Control. 2019 Jan-Dec;26(1):1073274819864111. doi: 10.1177/1073274819864111. PMID 31317770